CLINICAL TRIAL: NCT05885594
Title: Imaging Inflammation in Individuals With Alcohol Use Disorder: an [18F]NOS Study
Brief Title: Imaging Inflammation With Alcohol Use Disorder: an [18F]NOS Study
Acronym: AUD
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 851462
Record Dates: First submitted 2023-05-08; First posted 2023-06-02 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Use; Healthy Volunteer
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — Fluorine-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AUD-Alcohol Use Disorder (Other): 60 adult men and women who have alcohol use disorder will undergo up to 2 PET/CT scans each approximately 60 minutes of dynamic scanning starting at the time of injection of [18F]NOS. PET/CT imaging sessions will include an injection of ≤ 6.5 mCi (approximate range for most studies is anticipated to be 3.5-6.5 mCi) of [18F]NOS.
  Interventions: Drug: [18F]NOS
- HV-Healthy Volunteer (Other): 30 adult men and women between the ages of 18-65 who do not have alcohol use disorder and are a healthy volunteer will be enrolled in this study.
  Interventions: Drug: [18F]NOS

INTERVENTIONS:
Drug: [18F]NOS — [18F]-6-(2-fluoro-propyl)-4-methylpyridin-2-amine, also known as [18F]NOS, is a positron emitting radiopharmaceutical that has been studied in animals and humans which permits the visualization and measurement by positron emission tomography (PET/CT) imaging of in vivo iNOS expression as a marker of inflammation.
  Other Names: FNOS

SUMMARY:
Study to enroll up to 90 individuals, those with an alcohol use disorder (AUD) (up to n=60) and non-dependent healthy volunteers (HV) (up to n=30).

PET/CT imaging will be used to evaluate brain and whole-body inflammation using the investigational radiotracer [18F]NOS.

All participants will have one [18F]NOS positron emission tomography/ computed tomography (PET/CT) scan performed.

DETAILED DESCRIPTION:
The Investigators plan to enroll up to 90 individuals in this study, which will enroll individuals with an alcohol use disorder (AUD) (up to n=60) and non-dependent healthy volunteers (HV) (up to n=30).

PET/CT imaging will be used to evaluate brain and whole-body inflammation using the investigational radiotracer [18F]NOS. All participants will have one [18F]NOS positron emission tomography/computed tomography (PET/CT) scan performed, unless this has been performed as part of another study. AUD participants enrolled in a companion treatment study #851593 "A Randomized, Double-blind Placebo-Controlled Study of Ibudilast for Treating Alcohol Use Disorder" will be asked to undergo a second [18F]NOS PET scan after the initiation of the study treatment.

For each PET/CT scan, patients will undergo approximately 60 minutes of dynamic scanning starting at the time of injection of [18F]NOS. PET/CT imaging sessions will include an injection of ≤ 6.5 mCi (approximate range for most studies is anticipated to be 3.5-6.5 mCi) of [18F]NOS. Data will be collected to evaluate uptake of [18F]NOS in the brain and other organs (e.g., lungs, heart, and liver), and measurements will be compared between groups.

Each participant will undergo a 90 minute brain MRI to measure brain inflammatory markers using GluCEST and spectroscopic imaging, unless this has been performed as part of another study and deemed acceptable by an investigator. On the PET day, a blood sample will be collected to measure established peripheral inflammatory biomarkers to be correlated with [18F]NOS uptake. AUD participants who are enrolled in the companion treatment study will be asked to undergo a second brain MRI, PET/CT scan, and blood draw for inflammatory markers after the initiation of treatment.

ELIGIBILITY:
Inclusion Criteria for both study groups (AUD and HV)

* Age 18 years to 65 years old (inclusive)
* Willingness to provide signed informed consent and commit to completing the procedures in the study

Inclusion criteria for the AUD group:

* Meets DSM-5 criteria for AUD
* Average weekly ethanol consumption of at least 15 standard drinks over the past month prior to consent (self-report)
* Minimum 1 year history of heavy drinking (self-report).
* Must have had last drink within 1 week of the first PET visit.
* Alcohol specified as the preferred drug (self-report)
* Participants must agree to not consume alcohol beverages for 12 hours prior to laboratory sessions (self-report with 0 breath alcohol level)

Inclusion criteria for the AUD treatment group:

* Enrolled in the clinical trial titled "A Randomized, Double-blind Placebo-Controlled Study of Ibudilast for Treating Alcohol Use Disorder" and eliglible to be randomized into the study to receive study medication.

Inclusion criteria for the HV group:

* AUDIT score < 6
* Drinks alcohol 15 standard drinks or less per month (by self-report).

Exclusion Criteria for both study groups:

* Females who have a positive urine pregnancy test or are breast feeding at the time of screening will not be eligible for this study; a urine pregnancy test will be performed in women of child-bearing potential at screening, MRI, and at the PET/CT scan visits
* Current untreated and unstable diagnosis of substance use disorder that could interfere with study participation or make it hazardous for the subject to participate (except for nicotine or cannabis use disorder, and alcohol use disorder in the alcohol group)
* Positive urine drug screen for opiates, methamphetamine or cocaine at screening or study visit (may be repeated once and if result is negative on repeat it is not exclusionary)
* Individuals who are HIV positive, as the human immunodeficiency virus affects neurocognitive function, even in otherwise asymptomatic individuals, which can confound the results of PET and MRI testing
* Current, serious psychiatric illness (i.e., schizophrenia, bipolar disorder, psychotic major depression, panic disorder, or imminent suicide or violence risk) that could compromise participant safety or successful participation in the study
* Use of inhaled or oral corticosteroids or anti-inflammatory medications per medical record review or self-report and judged by a physician investigator to be potentially confounding
* Head trauma with loss of consciousness for more than 30 minutes or associated with skull fracture or inter-cranial bleeding or abnormal MRI (self-report, medical history)
* Presence of ferromagnetic objects in the body that are contraindicated for MRI of the head, fear of enclosed spaces, or other standard contraindication to MRI and or PET scanner (self-report checklist)
* Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
* Any current or past medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study
* Judged by the principal investigator or his designee to be an unsuitable candidate for study participation

Exclusion criteria for the HV group:

* Current DSM-5 diagnosis of Alcohol use disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
[18F]NOS uptake (distribution volume) in the brain and other organs in body | 2 hours
  The primary outcome measure to be analyzed is a comparisons of AUD subjects and healthy control subjects in the amount of [18F]NOS uptake (distribution volume) in brain and heart.

SECONDARY OUTCOMES:
Amount of c-reactive protein (mg/dl) in blood | 1 hour
  The secondary outcome measure is the comparison of AUD subjects and healthy control subjects in the amount of c-reactive protein in mg/dl, and its association with [18F]NOS uptake (distribution volume) in brain and other organs in body.
Amount of magnetic resonance spectroscopy Glutamate levels (in mM) in the brain | 1 hour
  The third outcome measure to be analyzed is the comparison of AUD subjects and healthy control subjects in brain Glutamate levels (in mM), and its association with [18F]NOS uptake (distribution volume) in brain.

OTHER OUTCOMES:
[18F]NOS uptake (distribution volume) in the brain and other organs in body pre and post treatment with Ibudilast | 2 hours
  The fourth outcome measure to be analyzed is a comparisons the amount of [18F]NOS uptake (distribution volume) in brain other organs pre and post 3-6 weeks treatment with Ibudilast for AUD.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Dubroff, MD, PhD, Principal Investigator — Perelman School of Medicine, Dept. of Radiology
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No